CLINICAL TRIAL: NCT03646266
Title: Partial Neuromuscular Blockade to Facilitate Lung and Diaphragm Protective Mechanical Ventilation in Intensive Care Unit Patients: a Randomized Controlled Pilot Study
Brief Title: Partial Neuromuscular Blockade for Lung Protective Mechanical Ventilation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Diana Jansen, Collaborating investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL65192.029.18
Record Dates: First submitted 2018-07-26; First posted 2018-08-24 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Rocuronium

STUDY DESIGN:
Intervention Model Description: pilot randomized controlled trial (RCT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rocuronium (Experimental): Titration of rocuronium bromide until tidal volume of 6ml/kg predicted body weight (PBW) is reached
  Interventions: Drug: Rocuronium Bromide
- Control (No Intervention): Standard of care

INTERVENTIONS:
Drug: Rocuronium Bromide — Titration with rocuronium bromide until tidal volume 6ml/kg PBW
  Other Names: Esmeron
  Arms: Rocuronium

SUMMARY:
Controlled mechanical ventilation may lead to the development of diaphragm muscle atrophy, which is associated with weakness and adverse clinical outcome. Therefore, it seems reasonable to switch to partially supported ventilator modes as soon as possible. However, in patients with high respiratory drive, the application of partially supported modes may result in high lung distending pressures and diaphragm injury.

Recently, the investigators published a study that demonstrated that a low dose of neuromuscular blocking agents (NMBA) facilitates lung-protective ventilation and maintains diaphragm activity in intensive care unit (ICU) patients. That study was conducted in a small (N=10), selected group of patients and partial neuromuscular blockade was applied for only 2 hours (proof-of-concept study). Therefore, further research has to be done before this strategy can be applied in clinical practice.

The primary goal is to investigate the feasibility and safety of prolonged (24 hours) partial neuromuscular blockade in patients with high respiratory drive in partially supported mode. The secondary goals are to evaluate the effect of this strategy diaphragm function, lung injury, hemodynamics and systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* high respiratory drive, defined as tidal volume > 8ml/kg PBW on inspiratory support of 12 cmH2O.
* sedation level: richmond agitation-sedation scale (RASS) ≤ -3
* ventilated in pressure support mode

Exclusion Criteria:

* recent use of NMBA (< 2 hrs)
* arterial pH < 7.25
* hemodynamic instability, i.e. high dose vasopressors (>0.5 μg/kg/min) or inotropes (dobutamine >15 μg/kg/min or enoximone >25 μg/kg/min)
* intracranial pressure > 20 cmH2O
* past medical history of neuromuscular disorders
* known pregnancy
* known previous anaphylactic reaction to NMBA's.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of breaths with tidal volume 6ml/kg predicted body weight (PBW) | At five time points of 1hr during the first 24hrs of the study period
  During the study period we measure at five time points of 1 hour (T0, T1, T5, T12, T24) all breaths and determine the percentage of breaths with a tidal volume of 6ml/kg PBW.
Incidence of directly related serious adverse events | During the 48hrs study period
  A serious adverse event is any untoward medical occurence or effect that:
  * results in death
  * is life threatening
  * requires prolongation of existing inpatients' hospitalization
  * results in persistent or significatn disability or incapacity
  * is a new event of the trial medication to affect the safety of the subjects, such as adverse events which are not already were described

SECONDARY OUTCOMES:
Number of patients completing the study without meeting the stopping criteria | At four time points during the first 24hrs of the study period
  After each time point (T0, T1, T5 and T12) we screen if the patient meets one of the stopping criteria, defined as:
  * potential of hydrogen (pH) < 7.20
  * heart rate > 100 beats per minute or an increase of > 20% from baseline for more than 20 minutes
  * increase in mean arterial blood pressure of > 20% for more than 20 minutes
Effect on partial carbon dioxide (pCO2) | During the 48hrs study period
  At three time points (T0, T24, T48) during the study period we will collect a blood sample from the arterial catheter, to measure the effect of prolonged NMB administration on pCO2 (in kPa), in order to:
  * determine if there were differences between the start and end of the study period
  * investigate if there were differences between both study groups
Effect on pH | During the 48hrs study period
  At three time points (T0, T24, T48) during the study period we will collect a blood sample from the arterial catheter, to measure the effect of prolonged NMB administration on pH, in order to:
  * determine if there were differences between the start and end of the study period
  * investigate if there were differences between both study groups.
Effect on heart rate | During the 48hrs study period
  During the study period we will collect at six time points (T0, T1, T5, T12, T24 and T48) the heart rate (in beats per minute), in order to:
  * determine if there were differences between the start and end of the study period
  * investigate if there were differences between both study groups.
Effect on blood pressure | During the 48hrs study period
  During the study period we will collect at six time points (T0, T1, T5, T12, T24 and T48) the blood pressure (millimetre(s) of mercury (mmHg)), in order to:
  * determine if there were differences between the start and end of the study period
  * investigate if there were differences between both study groups.
Effect on respiratory rate | During the 48hrs study period
  During the study period we will collect at six time points (T0, T1, T5, T12, T24 and T48) the respiratory rate (in breaths per minute) in order to:
  * determine if there were differences between the start and end of the study period
  * investigate if there were differences between both study groups.
Effect on peripheral capillary oxygen saturation (SpO2) | During the 48hrs study period
  During the study period we will collect at six time points (T0, T1, T5, T12, T24 and T48) the SpO2 (%) in order to:
  * determine if there were differences between the start and end of the study period
  * investigate if there were differences between both study groups.
Effect on partial oxygen pressure (pO2) | During the 48hrs study period
  At three time points (T0, T24, T48) during the study period we will collect a blood sample from the arterial catheter, to measure the effect of prolonged NMB administration on pO2 (in kPa), in order to:
  * determine if there were differences between the start and end of the study period
  * investigate if there were differences between both study groups.
Effect on work of breathing (WOB) | During the first 24hrs of the study period
  During the study period we will collect at five time points (T0, T1, T5, T12 and T24) the WOB (in Joule) in order to:
  * determine if there were differences between the start and end of the study period
  * investigate if there were differences between both study groups.
Effect on pressure time product (PTP) | During the first 24hrs of the study period
  During the study period we will collect at five time points (T0, T1, T5, T12 and T24) the PTP (in cmH2O per second) in order to:
  * determine if there were differences between the start and end of the study period
  * investigate if there were differences between both study groups.
Effect on tumor necrosis factor (TNF)-alfa | During the first 24hrs of the study period
  At three time points (T0, T24, T48) during the study period we will collect a blood sample from the arterial catheter, to measure the effect of prolonged NMB administration on TNF-alfa concentration (in pg/ml), in order to:
  * determine if there were differences between the start and end of the study period
  * investigate if there were differences between both study groups.
Effect on interleukin(IL)-6 and IL-8 | During the first 24hrs of the study period
  At three time points (T0, T24, T48) during the study period we will collect a blood sample from the arterial catheter, to measure the effect of prolonged NMB administration on IL-6 and IL-8 concentration (in pg/ml), in order to:
  * determine if there were differences between the start and end of the study period
  * investigate if there were differences between both study groups.
Amount of days on mechanical ventilation | Until 30 days after the end of the study period
  After 30 days we will investigate if there were differences between both groups in the duration of mechanical ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided